CLINICAL TRIAL: NCT02374749
Title: COmorbidities and EDucation in SpondyloArthritis Study (COMEDSPA) Evaluation of Standardized Follow-up in Axial Spondyloarthritis
Brief Title: COMorbidities and EDucation in SPondyloArthritis Study
Acronym: COMEDSPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P140401
Record Dates: First submitted 2015-01-01; First posted 2015-03-02 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Axial Spondyloarthritis
Keywords: Axial Spondyloarthritis; Education; Co-morbidities; Nurse
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — Comorbidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- comorbidities (Active Comparator): Evaluation of the prevalence and the presence of the risks factors of the four most frequently observed comorbidities in spondyloarthritis (cardiovascular diseases, cancers, infections osteoporosis and gastro-intestinal) as it is recommended by the French Society of Rheumatology.
  Interventions: Behavioral: Comorbidities (detection/prevention)
- self-assessment (Active Comparator): During the initial visit, the clinical research nurse exempt a learning program of assessment of disease activity/severity :
  * for assessing the activity in SpA;
  * for the calculation of BASDAI and the ASDAS-CRP
  * for the transfer technique and for the calculation of the disease activity on a monthly basis during the next 12 months.
  * for the risk of tobacco exposure
  * for the benefit of an NSAID intake in case of painful episode of the disease
  * for the benefit of home exercises
  * for the spine and indication of a treatment under the supervision of a physiotherapist in case of severe disease
  * for learning the patient to calculate his BASDAI and ASDAS-CRP Then, the patient will return home with his calculator and his notebook. Each month, the patient will be asked to perform the BASDAI and ASDAS-CRP calculations and to report the data on the notebook. 12 months later, the patient comes for a visit in the current practice to assess both such program and comorbidities.
  Interventions: Behavioral: self-assessment/self-management

INTERVENTIONS:
Behavioral: self-assessment/self-management — Nurse led-program of self-assessment/ self-management of spondyloarthritis
  Arms: self-assessment
Behavioral: Comorbidities (detection/prevention) — Standardized assessment of comorbidities by nurses
  Arms: comorbidities

SUMMARY:
Giving both the gap existing between the current recommendations to prevent/detect comorbidities and the clinical practice in patients suffering from spondyloarthritis and also the specificity of some recommendations to rheumatic diseases, it seems logical to check these recommendations in a rheumatologic "environment".

This study with its two parts should be able to demonstrate:

* The importance of a systematic evaluation of comorbidities in Spondyloarthritis,
* The utility of a nurse-led program of self-assessment and self-management of the disease

DETAILED DESCRIPTION:
Patients with spondyloarthritis will be invited by their rheumatologists to participate at this study in 21 centers in France.

500 patients are planned to be included.

After written informed consent will be obtained, the patients will be randomized in two arms:

* comorbidities
* self-assessment/self-management The patients will be seen again in the same center 12 months later in order to collect the outcome measures

The two primary objectives of this trial are :

* To evaluate the impact of a nurse led program of self-assessment of disease activity/severity and self-management on the level of satisfaction/coping
* To evaluate the impact of a nurse led program of assessment of comorbidities on the management of such comorbidities

The Secondary objectives are:

* To evaluate the prevalence of comorbidities in SpA;
* To evaluate the level of adherence to recommendations of prevention of comorbidities;
* To evaluate the impact of the nurse led program of self-assessment / self-management on the amount of NSAID (Non-steroidal Anti-Inflammatory Drugs) intake and the level of disability (e.g. functional disability)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female over 18 and under 80 years
2. Axial Spondyloarthritis according to the ASAS criteria (Assessment of SpondyloArthritis international Society)
3. Disease duration of at least one year
4. Activity of SpA to be stable according to the treating rheumatologist for at least three months before the date of inclusion
5. Lack of elective surgery during the 6 months after inclusion
6. Able to understand and adhere to the study treatments
7. Development of a medical examination results given to the patient
8. Informed Consent signed and dated

Exclusion Criteria:

1. Pregnant women (any method of contraception will be accepted)
2. Patients who have had a change in the treatment of SpA during the 3 months prior to inclusion
3. History of alcoholism, drug addiction, psychological problems, severe comorbidities that could possibly invalidate informed consent or limit patient compliance with the study protocol
4. No affiliation to a social security regime

   -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2017-10-16 (Actual)

PRIMARY OUTCOMES:
Comorbidities | 1 year later
  Changes after 12 months in the comorbidity composite score. Such composite score has been established prior the study and is taking into account the optimal management of patients (e.g. Normal blood pressure, no smoking,....) . Such score will be calculated at baseline and at the one year visit in the two groups.
self-assessment/self-management | 1 year later
  The level of coping after 12 months based on the question#8 ( 0-10 NRS) of the RAID score. Such outcome will be evaluated at both the baseline and the one year visits in both groups.

SECONDARY OUTCOMES:
Frequency of comorbidities in Spondyloarthritis | 1 year later
  This analysis will be purely descriptive and will include the percentage of patients with:
  * History of cardiovascular diseases
  * Hypertension
  * Diabetes
  * Hyperlipidemia
  * History of skin cancer, colon, uterus, breast, prostate
  * Percentage of patients at high risk of cancers when these risks are known (eg, family history of breast cancer, colon)
  * History of tuberculosis, HIV, or hospitalization for severe infections.
Frequency of compliance with general recommendations on vaccinations, screening for certain cancers and osteoporosis screening | 1 year later
  The percentage of patients adhering to these recommendations will be assessed.
Impact of self-assessment by the patient of his/her Spondyloarthritis activity (ASDAS-CRP (C Reactive Protein), BASDAI) on the activity and severity of the disease | 1 year later
  The final value of BASDAI and ASDAS-CRP will be compared in the two groups of patients by adjusting the analysis of the initial value.
  The final visit BASFI value will be compared in the two groups of patients by adjusting the analysis of the initial value
Patient compliance program self-management of Spondyloarthritis | 1 year later
  Compliance will be assessed by the percentage of the collections of the disease activity (BASDAI, ASDAS-CRP) actually made by the patient with regard the theoretical number one (e.g. monthly).

CONTACTS AND LOCATIONS:
Overall Officials: Maxime DOUGADOS, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Cochin, Paris, France

REFERENCES:
- [Background] Molto A, Gossec L, Poiraudeau S, Claudepierre P, Soubrier M, Fayet F, Wendling D, Gaudin P, Dernis E, Guis S, Pouplin S, Ruyssen-Witrand A, Chales G, Mariette X, Beauvais C, Combe B, Flipo RM, Richette P, Chary-Valckenaere I, Saraux A, Sibilia J, Schaeverbeke T, Dougados M. Evaluation of the impact of a nurse-led program of patient self-assessment and self-management in axial spondyloarthritis: results of a prospective, multicentre, randomized, controlled trial (COMEDSPA). Rheumatology (Oxford). 2021 Feb 1;60(2):888-895. doi: 10.1093/rheumatology/keaa480. PMID 33063096
- [Background] Molto A, Gossec L, Poiraudeau S, Claudepierre P, Soubrier M, Fayet F, Wendling D, Gaudin P, Dernis E, Guis S, Pouplin S, Ruyssen A, Chales G, Mariette X, Beauvais C, Combe B, Flipo RM, Richette P, Chary-Valckenaere I, Saraux A, Sibilia J, Schaeverbeke T, Dougados M. Evaluation of the impact of a nurse-led program of systematic screening of comorbidities in patients with axial spondyloarthritis: The results of the COMEDSPA prospective, controlled, one year randomized trial. Semin Arthritis Rheum. 2020 Aug;50(4):701-708. doi: 10.1016/j.semarthrit.2020.05.012. Epub 2020 May 27. PMID 32521324